CLINICAL TRIAL: NCT04631055
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of Intracranial Drug-coated Balloon Catheters in the Treatment of Symptomatic Intracranial Atherosclerotic Stenosis
Brief Title: AcoArt sICAS: DCB in the Treatment of Symptomatic Intracranial Atherosclerotic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AcoArt sICAS
Record Dates: First submitted 2020-11-03; First posted 2020-11-17 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Intracranial Atherosclerosis; Stroke
Keywords: Intracranial Atherosclerosis; Stroke; drug coated balloon
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB group (Experimental): use intracranial drug coated balloon catheter made by Acotec Scientific Co.,Ltd.
  Interventions: Device: drug coated balloon
- Stent group (Active Comparator): use the Intracranial Stent System made by MicroPort.
  Interventions: Device: stent system

INTERVENTIONS:
Device: drug coated balloon — paclitaxel coated balloon catheter for intracranial PTA treatment
  Arms: DCB group
Device: stent system — The Intracranial Stent System comprises of a balloon expandable stent and a delivery catheter that features a rapid exchange catheter design with a semi-compliant balloon located at its distal end.The product, APOLLO™ stent system, has the indication of endovascular treatment for intracranial stenosis approved by NMPA.
  Arms: Stent group

SUMMARY:
The purpose of the RCT trial is to determine whether DCB is not inferior to stent in treating intracranial stenosis.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, 1:1 randomized using paclitaxel coated balloon versus stent to treat intracranial stenosis of 70-99% degree. And primary endpoint is angiographic restenosis at 6 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age;
* Patients with symptomatic intracranial atherosclerotic stenosis;
* Patients with intracranial arterial de novo stenosis confirmed by digital subtraction angiography (DSA);
* Confirmed by DSA，the diameter of the target vessel is between 2.5mm-4.5mm ; according to WASID method, the degree of stenosis of the target lesion is 70%-99%;
* Baseline mRS score ≤2;
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients with stroke within 2 weeks before procedure;
* Patients with stroke caused by perforating artery occlusion;
* Any history of brain parenchymal or other intracranial subarachnoid, subdural or extradural hemorrhage in the past 30 days;
* Those who have received thrombolysis within 24 hours before procedure;
* Deterioration of neurological function within 24 hours before procedure (defined as NIHSS score increased by ≥ 4 points over the baseline);
* The vascular path showed in angiography is so tortuous that it is difficult to advance catheters to the target lesion or retrieve;
* Lesions that investigators believe are not suitable for stenting;
* Patients with thrombus in target vessel;
* In addition to the target lesion, there are still other de novo lesion or ISR lesion with more than 70% diameter stenosis in intracranial arteries that need to be treated at the same time;
* After endovascular treatment of the target lesion, there is still a stenosis of more than 50% in the main blood supplying artery or an obstructive lesion in the distal vessel of target lesion;
* Major surgery (including open femoral artery, aortic or carotid artery surgery) within the past 30 days or planned within 90 days;
* Patients with renal artery, iliac artery, and coronary artery requiring simultaneous intervention;
* Combined with intracranial tumor, aneurysm or intracranial arteriovenous malformation;
* Intracranial artery stenosis caused by non-atherosclerotic lesions, including: arterial dissection, moya-moya disease, vasculitis disease, herpes zoster, varicella-zoster or other viral vascular diseases, neurosyphilis, any Other intracranial infections, any intracranial stenosis related to cerebrospinal fluid cells, radiation-induced vascular disease, fibromuscular dysplasia, sickle cell disease, neurofibromatosis, central nervous system benign vascular disease, postpartum vascular disease, suspected Vasospasm, suspicious embolism recanalization, etc.;
* Cardiac stroke or potential cardiogenic thromboembolism, with any of the following cardiogenic embolism causes: chronic or paroxysmal atrial fibrillation, mitral valve stenosis, mechanical valves, endocarditis, intracardiac thrombus or implant, dilated cardiomyopathy, spontaneous acoustic imaging of the left atrium;
* Patients with myocardial infarction within 6 weeks before procedure;
* Those who cannot tolerate general anesthesia due to insufficiency of important organs such as heart and lungs;
* Patients with known severe hepatic and renal dysfunction;
* Patients with hemoglobin<100g/L, platelet count<100×1,000,000,000/L, INR>1.5 or there are uncorrectable factors leading to bleeding(if there are multiple checks, the last one shall prevail);
* Patients who cannot receive dual antiplatelet therapy due to existing diseases or are tolerant to dual antiplatelet therapy confirmed by relevant test;
* Patients with known severe allergies or contraindications to heparin, paclitaxel, contrast agents and other related intravascular treatment drugs;
* Current alcohol or drug abuse, uncontrolled severe hypertension (systolic blood pressure>180mmHg or diastolic blood pressure>110mmHg);
* Life expectancy <1 year;
* Pregnant or lactating women;
* Patients who cannot complete the follow-up due to cognitive, emotional or mental illness;
* Patients who are participating in other drug/device clinical trials and have not completed all follow-ups required by the programmer;
* According to the judgement of the investigator, other situations that are not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Angiographic restenosis of the target lesion | 6 months post-procedure
  Definition of Restenosis:
  1. Post-procedural residual stenosis < 30% of target lesion occurs >50% stenosis within the treated segment at 6 months angiographic follow-up.
  2. Post-procedural residual stenosis 30-50% of target lesion occurs >20% absolute luminal loss within the treated segment at 6 months angiographic follow-up.
Primary safety endpoint: Target vessel stroke or death event | within 30 days post-procedure
  Stroke (Hemorrhagic stroke and ischemic stroke) or death related to target vessels within 30 days postoperatively.

SECONDARY OUTCOMES:
Device success rate | during procedure
  DCB: The balloon dilatation catheter was able to reach the treated lesion, successfully dilated without rupture, and successfully retreated.
  Stent: Successful delivery and deployment of the stent and the delivery system of stent could be retreated successfully.
Target vessel ischemia stroke event | between 31 days and 6 months post-procedure
  The incidence of recurrent ischemic stroke in the target vessel supply area 31 days to 6 months postoperatively
Cerebral parenchyma hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage events | between 31 days and 6 months post-procedure
  Any parenchymal hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage 31 days to 6 months postoperatively
Target vessel death event | between 31 days and 6 months post-procedure
  Target-vessel related death 31 days to 6 months postoperatively
Transient ischemic attack event | at 6 months post-procedure
  transient ischemic attack event transient ischemic attack event
National Institutes of Health Stroke Scale score | at 6 months post-procedure
  National Institutes of Health Stroke Scale score at 6 months post-procedure(0-42,higher scores mean a worse outcome)
Modified Rankin Scale score | at 6 months post-procedure
  Modified Rankin Scale score at 6 months post-procedure(0-5,higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Beijing
  - Nanyang City Central Hospital, Nanyang
  - Shanxi Cardiovascular Hospital, Taiyuan

REFERENCES:
- [Derived] Ma G, Sun D, Jia B, Ling L, Nguyen TN, Sun X, Yu B, Wen C, Cheng T, Chen W, Han J, Han H, Guo G, Yu J, Wei L, Huang R, Mao G, Shen Q, Yang X, Wang B, Luo G, Huo X, Gao F, Mo D, Ma N, Miao Z. Comparison of drug-coated balloon with bare-metal stent in patients with symptomatic intracranial atherosclerotic stenosis: the AcoArt sICAS randomized clinical trial. J Neurointerv Surg. 2025 Feb 25:jnis-2024-022768. doi: 10.1136/jnis-2024-022768. Online ahead of print. PMID 40010849